CLINICAL TRIAL: NCT03985618
Title: The MODE Trial: A Pilot Trial Investigating Planned Caesarean Section Versus Induction of Labour for Women With Class III Obesity
Brief Title: The MODE Trial: Planned Caesarean Section Versus Induction of Labour for Women With Class III Obesity
Acronym: MODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRRF ID 1469; FDN148438 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2019-05-21; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Obesity Complicating Childbirth; Obesity; Labor Onset and Length Abnormalities; Pregnancy, High Risk; Cesarean Section Complications
Keywords: obesity; pregnancy; labour; labor; caesarean; cesarean; C-section; induction
MeSH Terms: conditions — Obesity | interventions — Cesarean Section; Labor, Induced

STUDY DESIGN:
Intervention Model Description: Brewin partially randomized control trial, patient preference trial. In this design, each eligible patient is asked for her preference for mode of delivery. Patients with a preference are given their delivery mode of choice. If a patient does not have a preference, randomization takes place. Advantages to this design include the fact that preferences are taken into account in care allocation and that almost all those who are eligible enter the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized Caesarean section (Active Comparator): Randomized to planned pre-labour Caesarean section
  Interventions: Procedure: Caesarean section
- Randomized Induction of Labour (Active Comparator): Randomized to planned induction of labour
  Interventions: Procedure: Induction of Labour
- Preference Caesarean section (Active Comparator): Preference for planned pre-labour Caesarean section
  Interventions: Procedure: Caesarean section
- Preference Induction of Labour (Active Comparator): Preference for planned Induction of Labour
  Interventions: Procedure: Induction of Labour

INTERVENTIONS:
Procedure: Caesarean section — Planned pre-labour Caesarean section at 38-40 weeks. For patients planning Caesarean Section, surgical planning, precise timing and method of Caesarean section is at the discretion of the most responsible care provider, as per local procedures.
  Other Names: C-section; Cesarean
  Arms: Preference Caesarean section; Randomized Caesarean section
Procedure: Induction of Labour — Planned induction of labour at 38-40 weeks. For patients planning induction of labour, precise timing and method of induction of labour is at the discretion of the most responsible care provider, as per local procedures.
  Arms: Preference Induction of Labour; Randomized Induction of Labour

SUMMARY:
Canadian guidelines recommend that women with a pre-pregnancy body mass index (BMI) at or above 40 kg/m2 deliver by their due date. When delivery is planned prior to spontaneous labour, there are two options: planned induction of labour or pre-labour Caesarean (C-section). However, it is not yet clear whether induction of labour or planned pre-labour C-section is the best option for this population.

The MODE Trial aims to assess the feasibility of conducting a larger-scale trial of planned mode of delivery in first time mothers who have a BMI >=40kg/m2, and obtain preliminary data on health outcomes for moms and babies following delivery by either planned C-section or induction of labour.

DETAILED DESCRIPTION:
Women with obesity have a decreased likelihood of achieving vaginal delivery. According to the Centre for Maternal and Child Enquiries, the chance of spontaneous vaginal delivery in women with a BMI ≥35kg/m2 is 55%, while the chance is 36.7% in women with a BMI ≥40.0kg/m2. This number includes women who go into labour spontaneously, in which, the odds of a vaginal delivery are highest. The rate of failure to induce labour approaches 80% with increased complications and morbidity including abnormal fetal heart rate monitoring, labour dystocia, emergency C-section, and fetal macrosomia. It has been proposed that some women may benefit from a planned Caesarean section delivery. However, Caesarean sections are also not straightforward in women with obesity, and come with significant risks of short- and long-term morbidity for mother and baby, including prolonged operative times, higher volumes of blood loss and infection rates and higher rates of NICU admission.

Given that there are many considerations when deciding how to best deliver a woman with obesity, it is not surprising that there is a high degree of clinical equipoise. In reality, the decision is made jointly between the patient and her care provider, often guided by overall instinct and local resource availability.

Studies to date have been retrospective in nature. There is a significant need for prospective study of the outcomes and experiences of planned induction of labour and planned Caesarean section in women with obesity to allow evidence-based counselling and decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Capability of participant to comprehend and comply with study requirements
* Age ≥18 years at time of consent
* Nulliparous (never given birth after 19+6/7 weeks of gestation)
* Pre-pregnancy BMI or calculated BMI obtained in the first 13 weeks of pregnancy ≥40kg/ m2
* Participant plans to give birth in a participating site
* Gestational age 34+0/7 - 36+6/7 weeks (based on estimated date of conception (EDC) assigned at the first ultrasound performed after 7+0/7 and prior to 20 +0/7 weeks)
* Live fetus, documented positive heart rate at visit 1 prior to randomization
* Singleton fetus in cephalic presentation at the time of randomization
* No maternal or fetal contraindications to vaginal delivery

Exclusion Criteria:

* Known major fetal anomaly, confirmed by ultrasound or genetic testing
* Multiple gestation
* Known documented evidence of alcohol or drug abuse in this current pregnancy
* Currently enrolled or has participated in another clinical trial within 3 months of the date of randomization (at discretion of Trial Coordinating Centre)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting a larger-scale trial (eligibility criteria) | 18 months
  Appropriateness of eligibility criteria, measured by the reasons for exclusion of screened patients
Feasibility of conducting a larger-scale trial (recruitment rate) | 18 months
  Eligibility and recruitment rate, measured by the proportion of patients who are eligible and recruited into the trial
Feasibility of conducting a larger-scale trial (randomization) | 18 months
  Appropriateness of randomization, measured by the proportion of trial participants who consent to randomization

SECONDARY OUTCOMES:
Maternal morbidity and mortality | Pregnancy to 6 week postpartum
  Rates of: maternal death, admission to ICU, intrapartum Caesarean section, postpartum hemorrhage, postpartum wound infection, endometritis, venous thromboembolism (VTE), hypertensive disorders of pregnancy (gestational hypertension or preeclampsia), indication for Caesarean delivery, operative vaginal delivery, indication for operative vaginal delivery, uterine incision extensions during Caesarean section, chorioamnionitis, third or fourth degree perineal lacerations, induction agents, pain medication use during induction, labour, Caesarean section and postpartum.
Fetal and neonatal morbidity and mortality | Pregnancy to 6 week postpartum
  Rates of: stillbirth, neonatal death, gestational age at birth, birthweight, need for respiratory support within 72 hours of birth, duration of respiratory support, 5 minute Apgar <7, hypoxic-ischemic encephalopathy, seizure, infection (confirmed sepsis or pneumonia), meconium aspiration syndrome, birth trauma (bone fracture, neurologic injury or retinal hemorrhage), cephalohematoma, intracranial or subgaleal hemorrhage, or hypotension requiring vasopressor support, breastfeeding rates, hypoglycemia requiring intravenous treatment, jaundice requiring treatment, need for transfusion.
Length of hospital stay | Start of induction to delivery; admission to delivery; and delivery until discharge, assessed up until 6-weeks postpartum
  Length of hospital stay (in minutes) for both mom and baby
Hospital readmission rates | Delivery to 6-weeks postpartum
  The proportion of mothers and/or infants re-admitted to the hospital
Techniques for induction of labour | Admission to hospital until delivery, assessed up to 7 days from hospital admission.
  What method was used for induction
Maternal satisfaction | Approximately 48-hours post-birth and 42+/-7 days postpartum
  Maternal satisfaction with study design and procedures, measured by a survey
Healthcare provider satisfaction | 18 months
  Healthcare provider satisfaction with study design and procedures, measured through a survey

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gaudet, MD, MSc, Principal Investigator — The Ottawa Hospital; Ruth Rennicks White, BScN, Study Director — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No